CLINICAL TRIAL: NCT00952536
Title: The Effect of Daily Dietary Intake of Dried Whole Food Concentrates of Fruit, Vegetables and Berries (Juice Plus+) in Improving Clinical Outcomes Following Non-surgical Periodontal Therapy: a Pilot Study.
Brief Title: Effect of Dietary Intake of Dried Whole Food Concentrates (Juice Plus) on Clinical Outcomes Following Periodontal Therapy: A Pilot Study
Acronym: BHAM-NSA-05-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Birmingham Community Healthcare NHS (Other Government)
Collaborators: NSA, LLC (Industry)
Responsible Party: Principal Investigator, Professor I Chapple, Professor (PI for study), Birmingham Community Healthcare NHS
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BHAM-NSA-05-001 vs 11
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Periodontitis
Keywords: Randomised controlled trial; Double blind fully masked; Dietary supplement
MeSH Terms: conditions — Periodontitis | interventions — Vegetables; Fruit; Farms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Triple therapy (Active Comparator): Daily Juice Plus+ with 2 vegetable & 2 fruit & 2 berry capsule (test group 1)
  Interventions: Dietary Supplement: Daily Juice Plus+ with vegetable & fruit & berry capsule
- Dual Therapy (Active Comparator): Juice Plus+ with 2 vegetable & 2 fruit & 2 placebo capsule (test group 2)
  Interventions: Dietary Supplement: Daily Juice Plus+ vegetable & fruit & placebo capsule
- Control (Placebo Comparator): Daily Placebo in the form of 6 capsules (control group)
  Interventions: Dietary Supplement: Placebo in the form of 6 capsules

INTERVENTIONS:
Dietary Supplement: Daily Juice Plus+ with vegetable & fruit & berry capsule — Daily Juice Plus+ with 2 vegetable & 2 fruit & 2 berry capsule
  Other Names: Daily Juice Plus+ Fruit, Vegetable and Vineyard
  Arms: Triple therapy
Dietary Supplement: Daily Juice Plus+ vegetable & fruit & placebo capsule — Daily Juice Plus+ with vegetable & fruit & placebo capsule
  Other Names: Juice Plus+ Vegetable & Fruit & placebo capsule
  Arms: Dual Therapy
Dietary Supplement: Placebo in the form of 6 capsules — Daily Placebo in the form of 6 capsules (control group)
  Other Names: Placebo
  Arms: Control

SUMMARY:
There are 3 hypotheses to be tested:

1. That daily supplementation with Juice Plus+ will significantly improve treatment outcomes over placebo supplementation, at 3-months post-therapy, when used as an adjunct to conventional non-surgical periodontal therapy.
2. Triple therapy with Juice Plus+ (fruit, vegetable & berry) will produce additional treatment benefit over dual therapy (fruit & vegetable) and over placebo.
3. Improved treatment outcomes with Juice Plus+ will be maintained at 9-months post-therapy.

Brief Summary:

Periodontal diseases are highly prevalent chronic inflammatory diseases and a major cause of tooth loss. Data supports an association between periodontitis prevalence and reduced serum levels of antioxidants. Anecdotal reports from periodontal specialists indicate significant improvements in clinical outcomes from periodontal therapy where adjunctive Juice Plus+ is used, in agreement with research data from other systemic diseases where hyper-inflammation is implicated in disease pathogenesis. There is however, a lack of scientific evidence from clinical trials of periodontitis. Given the demonstrable antioxidant deficiency in periodontitis patients (both locally and peripherally), the excess oxidative stress in periodontitis patients, and the anecdotal evidence of clinical benefit from the adjunctive use of Juice Plus+, this study proposes to investigate the impact of daily supplementation with Juice Plus+ as an adjunct to traditional non-surgical periodontal therapy, in improving therapeutic outcomes.

DETAILED DESCRIPTION:
This will be a longitudinal, randomised, stratified (for age), double-blind, 3-arm study of non-surgical periodontal therapy. The 3 arms will be:

1. Daily Juice Plus+ with 2 vegetable & 2 fruit & 2 berry capsule (test group 1)
2. Daily Juice Plus+ with 2 vegetable & 2 fruit & 2 placebo capsule (test group 2)
3. Daily Placebo in the form of 6 capsules (control group)

Volunteers will receive standard non-surgical periodontal therapy by a single operator (study hygienist) and outcome measures will be assessed at baseline, 3, 6 and 9-months post-therapy. Capsules will be taken with food twice daily (3 capsules am & 3 capsules pm).

60 non-smoking patients with chronic moderate/severe periodontitis will be recruited from outpatient periodontal clinics at Birmingham's Dental Hospital. Subjects will be 30-60 years of age, male or female. Chronic periodontitis (CP) will be defined as the presence of 2 or more sites per quadrant with pocketing or interproximal attachment loss of > 6mm and 1/3rd radiographic bone loss.

The following exclusion criteria will apply:

* Patients with aggressive disease
* Patients with physical or mental disability
* Pregnant women
* Patients whose medical history may place them at risk of complications from periodontal therapy (e.g. need for antibiotic cover, warfarinised subjects)
* Patients taking long term anti-microbial or anti-inflammatory drugs
* Patients unable to swallow Juice Plus+ capsules
* Patients unable to provide informed consent
* Current smokers
* Patients taking regular vitamin supplementation

Outcome measures Primary outcome measures of healing will be increases in attachment level and reductions in probing pocket depths at 3-months. In addition reduction in percentage sites bleeding on probing (BOP - measured dichotomously at 4 sites per tooth) from the marginal tissues and gingival redness assessed visually (Modified Gingival Index-MGI) will be used as a primary outcome measure of tissue inflammation.

Secondary outcome measures will be reduction in % sites with disclosed plaque (PS - measured dichotomously at 4 sites per tooth), reductions in gingival crevicular fluid (GCF) volume, increases in GCF and plasma TAOC.

Probing measures will be performed in duplicate with a constant force (UNC PC15) probe and where differences between duplicate measures of greater than 1mm arise, a 3rd measure will be taken. The mean of the two closest measures will be recorded. Mean probing attachment and pocket depth measures per subject will be calculated at each examination point (baseline, 3, 6 & 9-months post-therapy).

The bleeding and plaque scores will be expressed as means per subject at each examination point and MGI scores as % sites with codes 0, 1, 2 and 3 per subject.

Samples GCF samples will be collected (30s) using Periopaper strips from the mesio-buccal aspects of 3 deep (>6mm) and 3 shallow (<3mm) molar sites per subject as described in appendix 1. Volumes will be read on a pre-calibrated Periotron 8000 according to standard methodologies 19. Each trio of sample strips will be collected into 400ul PBS/BSA buffer and snap frozen under liquid nitrogen until assay 13.

Blood samples (2 x 7 mls) will be collected into Vacutainer™ tubes for plasma. Platelet depleted plasma will be prepared by centrifugation at 1000g for 30 mins (4C). Plasma will be aliquoted into cryogenic vials and half will be snap frozen under liquid nitrogen until TOAC assay. The remaining half will be aliquoted into two 1.5ml cryogenic vials and stored at -80C for future use (e.g. assay for carotenoid activity). All samples will be stored in the dark and kept free from direct sunlight at all stages of handling.

Enhanced chemiluminescent assay (ECL) for total antioxidant capacity (TAOC) The ECL assay for total AO capacity (TAOC) was developed by our group 12 and is based upon the horse radish peroxidase catalysed oxidation of luminol by hydrogen peroxide. A BioOrbit 1250 luminometer (Labtech International, Sussex, UK), interfaced with a PC running software which allows simultaneous recording / display of up to 5000 data points over a period up to 1 hour is used to quantify light output. The enhancer, p-iodophenol, is no longer commercially available but is synthesised "in house". Antioxidant capacities of test samples will be derived from standard curves produced using the water-soluble vitamin E analogue, 6-hydroxy-2,5,7,8, tetramethylchroman-2-carboxylic acid (Trolox; assay range: 0.0625-1.6 nanomole) which will be run before and after test samples and results expressed as a concentration (µM Trolox equivalents/L; Teq/L).

All samples from each subject throughout the study (n=12: 8 GCF's - comprising 1 pooled from deep sites & 1 pooled from shallow sites @ each of 4 visits & 4 plasma samples) will be assayed on the same day and under the same laboratory conditions, in duplicate (total = 24 per subject). Each day samples from a test group 1 subject, a test group 2 subject and a control subject will be run. All assays will be completed in 10-12 hours of laboratory time per day and over 20 laboratory days (72 assays per day & 36 standards = 108 assays per day).

GCF samples will be defrosted, eluted in running buffer for 30 minutes prior to assay, when 100ul aliquots will be assayed in duplicate. Plasma samples will be diluted 1:10 in PBS/BSA running buffer and assayed as 20ul aliquots in duplicate.

Calibrations will be run at the beginning, mid-point and end of each day.

Statistical Analysis This will be performed by an independent statistician appointed by National Safety Associates Inc. All three study hypotheses presume that two subjects with the same initial attachment level and pocket depth would have the same expected final attachment level and pocket depth, except for the effect of their respective treatments. Therefore, the first two hypotheses will be investigated by using Analysis of Covariance, with the 3 month value of attachment level or pocket depth as a response, initial value as a covariate, and treatment as a study factor. Hypothesis 3 will be investigated in a similar fashion, except that the response will be the 9-month measurement.

In order to test hypotheses 1 and 3, the Placebo group will be compared to the two active treatment groups combined. In order to test hypothesis 2, the two active treatment groups will be compared.

Graphical displays and regression models will be used to investigate whether response to the active treatments is related to a subject's fruit and vegetable intake as measured by the Visual Analogue Scale data.

Secondary outcomes will be analyzed in a similar fashion.

Both Intention-To-Treat (ITT) analyses and Per Protocol (PP) analyses will be performed. In the ITT analyses, the data from all subjects will be used, regardless of adherence to treatment. In the PP analyses, the statistical models will include measures of adherence.

All statistical tests will be two-sided and performed at the 0.05 level of significance. The analyses will be performed by using SAS for Windows, version 8.2 (SAS Institute Inc., Cary, NC, USA), and SYSTAT, version 10.2.01 (SYSTAT Software Inc., Point Richmond, CA, USA).

Missing data: The primary outcome measures are taken as part of standard care during the subjects' 9-month review. There is no reason for missing data to be related to treatment or outcome. We will check whether having missing data is related to treatment assignment, but otherwise expect to be able to ignore missing values in the analyses because they will be "missing completely at random".

Code Breaking The codes will be kept sealed and locked in the office of the PI and will not be broken until after the statistical analysis is complete.

Power Calculation As this is a pilot study it is not possible to perform a power calculation based upon antioxidant outcomes. However, using the primary outcome measure of reduction in probing pocket depth and assuming we can obtain additional PPD reductions of 0.5 mm (or 0.4mm) over non-surgical therapy alone through supplementation with Juice Plus+ capsules, then to have an 80% chance of finding a significant difference at the p<0.05 level we would need to exit 12 (or 17) patients per treatment. This is based on accepted mean PPD reductions for mild to moderate periodontal disease of 1-2mm with non-surgical therapy and data from a study we performed that demonstrated mean PPD reductions of 1.08 + 0.4mm (SD). Recruiting 20 per treatment and allowing for a drop out rate of 20% would still provide sufficient power.

Patient Adherence Adherence with taking supplementation will be checked at each visit during active therapy and again at the 3, 6, and 9-month visits. Subjects will be provided with a data sheet to log days when they have missed taking supplements. In addition, one cryogenic vial containing a minimum of 500ul plasma will be archived at baseline, 3, 6 and 9-months post-therapy for each subject and may be used for carotenoid assay for biochemical verification of adherence.

GCP Statement This study will be conducted in accordance with International Good Clinical Practice (GCP) standards.

Documentation and Record-keeping The investigator will retain and archive all documents and source (raw) data pertaining to the study for a minimum period of 10 years.

Clinical Study Report The interpretation of the data will be the joint responsibility of the Investigator and the study team. A final report will be made in writing and is the responsibility of the same group and will include:-

* appropriate statistical procedures,
* any deviation from the protocol;
* conclusions as to efficacy of the treatments and the significance of any differences between them.

ELIGIBILITY:
Inclusion Criteria:

* Chronic periodontitis
* Presence of 2 or more sites per quadrant with pocketing or interproximal attachment loss of greater than 6mm and 1/3rd radiographic bone loss

Exclusion Criteria:

* Subjects with aggressive disease
* Subjects with physical or mental disability
* Pregnant women
* Subjects whose medical history may place them at risk of complications from periodontal therapy (e.g. need for antibiotic cover, warfarinised subjects)
* Subjects taking long term anti-microbial or anti-inflammatory drugs
* Subjects unable to swallow Juice Plus+ capsules
* Subjects unable to provide informed consent
* Current smokers
* Subjects taking regular vitamin supplementation

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-02; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure of healing will be increases in attachment level and reduction in probing pocket depths at 3-months. | 3, 6 and 9-months

SECONDARY OUTCOMES:
Secondary outcome measures will be reduction in % sites with disclosed plaque (PS - measured dichotomously at 4 sites per tooth), reductions in gingival crevicular fluid (GCF) volume, increases in GCF and plasma TAOC. | 3, 6 and 9-months

CONTACTS AND LOCATIONS:
Overall Officials: Iain LC Chapple, BDS FDS PhD, Principal Investigator — The University of Birmingham
Locations (1):
- Birmingham Dental Hospital & Scool, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Chapple IL, Milward MR, Ling-Mountford N, Weston P, Carter K, Askey K, Dallal GE, De Spirt S, Sies H, Patel D, Matthews JB. Adjunctive daily supplementation with encapsulated fruit, vegetable and berry juice powder concentrates and clinical periodontal outcomes: a double-blind RCT. J Clin Periodontol. 2012 Jan;39(1):62-72. doi: 10.1111/j.1600-051X.2011.01793.x. Epub 2011 Oct 17. PMID 22093005